CLINICAL TRIAL: NCT04015830
Title: Exploring Racial Disparities in Sleep Health and Neurocognitive Function in Older Adults With HIV
Brief Title: Exploring Racial Disparities in Sleep Health and Neurocognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: UAB Resource Centers for Minority Aging Research (RCMAR) (Unknown)
Responsible Party: Principal Investigator, Shameka L. Cody, Assistant Professor, University of Alabama, Tuscaloosa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UATuscaloosa
Record Dates: First submitted 2019-04-29; First posted 2019-07-11 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: HIV Dementia
Keywords: Sleep; Neurocognitive Disorders; HIV/AIDS; Aging
MeSH Terms: conditions — AIDS Dementia Complex; Neurocognitive Disorders; Acquired Immunodeficiency Syndrome | interventions — Evoked Potentials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older Adults with HIV (N = 60) (Experimental): African Americans and Whites age 50 and older
  Interventions: Other: electroencephalography (EEG) and event related potentials (ERP)

INTERVENTIONS:
Other: electroencephalography (EEG) and event related potentials (ERP) — This is an exploratory study of EEG/ERP measures in older African American and Whites with HIV

SUMMARY:
Despite longer life expectancies due to combination antiretroviral therapy (cART), the prevalence of HIV-associated neurocognitive disorders (HAND) persists thus affecting 52% of the HIV population. Poor sleep quality is commonly reported in older adults and has been related to neurocognitive impairments. This is concerning given studies have shown that up to 75% of adults with HIV experience poor sleep, and by 2020, 70% of adults with HIV will be age 50 and older. It is important to examine sleep quality as it relates to neurocognitive function and HAND in older adults with HIV given its negative impact on cART adherence. Compared to Whites with HIV, African Americans (AA) are disproportionately affected by HIV and are more likely to experience poor sleep quality. This primary goal of this 1-year cross-sectional study is to examine racial differences in sleep quality and neurocognitive function among 60 African Americans and Whites with HIV (age 50+).

DETAILED DESCRIPTION:
This study is designed with two aims: Aim 1a: To explore differences in sleep health between older HIV+ AA and Whites. 1b: To explore differences in domain-specific neurocognitive impairments between older HIV+ AA and Whites. Aim 2a: To explore the relationship between sleep health and neurocognitive function. 2b: To explore the relationship between sleep health and cART adherence. 2c: To explore mediation effects of cART adherence between sleep health and neurocognitive function. This is the first study to explore racial disparities in sleep health and neurocognitive function, using EEG/ERP metrics, among older HIV+ adults. There are two phases in this study: Phase I which consists of neurocognitive testing and sleep assessments with actigraphy, and Phase II which consist of a 20-30 min EEG. Measurements of electrical brain activity will be captured while participants engage in an Attention Network Test which measures executive function, attention, and speed of processing.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Identify as AA or White
* 50 years old or older
* Speak English

Exclusion Criteria:

* Alzheimer's disease or dementia
* Severe neurocognitive impairment (>7 errors on the Short Portable Mental Status Questionnaire)
* Deaf or blind
* Currently undergoing radiation/chemotherapy
* Brain trauma with loss of consciousness greater than 30 minutes
* A learning disability
* Significant neuromedical comorbidities (e.g., schizophrenia)
* Currently taking Efavirenz
* Moderate to severe sleep apnea
* Restless leg syndrome
* Narcolepsy
* Left handedness

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Subjective Sleep Health | Day 1
  Pittsburgh Sleep Quality Index (PSQI), the components are summed to create a global score between 0 and 21, with a global score of 5 or greater indicating poor sleep quality
Sleep Onset and Wake Time | 7 days
  A sleep diary will be used to evaluate sleep onset and wake time. Participant will be asked to document the time they fall asleep and the time they wake up
Insomnia Severity | Day 1
  Insomnia Severity Index is a measure of insomnia. Total scores ranging from 0-28 with higher scores indicating more severe clinical insomnia
Speed of Processing | Day 1
  Trails Making A Test is a measure of speed of processing (timed task) with greater time to complete task (in minutes) indicating poorer speed of processing
Executive Function | Day 1
  Trails Making Test B is a measure of executive function (timed task) with greater time to complete task (in minutes) indicating poorer executive function
Attention | Day 1
  Paced Auditory Serial Addition Task is a measure of attention (50 items) with greater number of items correct indicating good attention span
Spatial Visualization | Day 1
  Wechsler Adult Intelligence Scale (WAIS III) is a measure of spatial visualization. Scores on items are summed for a maximum score of 21 with greater scores indicating better spatial visualization
Verbal Learning and Memory | Day 1
  Hopkins Verbal Learning Test-Revised (Recall and Delayed) is a measure of verbal learning and memory. Three learning trials are summed to calculate a total recall score (maximum score is 36) with greater scores indicating better verbal learning and memory. The delayed recall score is the number of items correct (maximum score is 12) after 25-minutes with greater scores indicating better delayed recall.
Brief Visuospatial Memory Test (BVMT) (Recall and Delayed) | Day 1
  Measure of visuospatial memory, three learning trials are summed to calculate a total recall score (maximum score is 36) with greater scores indicating better visuospatial memory. The delayed recall score is the number of items correct (maximum score is 12) after 25-minutes with greater scores indicating better delayed visuospatial memory.
Sleep Onset | Day 1
  Actigraphy will measure sleep onset which is the time (in minutes) it takes to fall asleep with longer times indicating worse sleep onset. Time (in minutes) is averaged over 7 days.
Total Sleep Time | Day 1
  Actigraphy will measure total sleep time which is the number of sleep hours with lesser hours indicating worse sleep deficiency. Time (in hours) is averaged over 7 days.
Wake After Sleep Onset | Day 1
  Actigraphy will measure wake after sleep onset which is the number of awakenings after sleep onset with greater number of episodes indicating sleep fragmentation/poorer sleep.
Sleep Efficiency | Day 1
  Actigraphy will measure sleep efficiency which is the percentage of time spent sleep while in bed. It is calculated by dividing the total sleep time (in minutes) by the total amount of time in bed (in minutes) with 85-95% indicating good sleep efficiency.
Reaction Time | Day 1
  The Attention Network Test is a computerized measure of reaction times (in milliseconds) to presented stimuli over several trials. Mean reaction time is calculated by averaging the reaction times over 7 trials, with longer mean reaction times indicating poorer attention.

SECONDARY OUTCOMES:
Medication Adherence | Day 1
  Simplified Medication Adherence Questionnaire is a measure of antiretroviral adherence, a participant is non-adherent if he/she has missed more than two doses within the last week or has not taken any medication for two complete days within the last three months
Instrumental Activities of Daily Living | Day 1
  Brody and Lawton Instrumental Activities of Daily Living is a measure of instrumental activities of daily living, scores from 8 categories (ability to use telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility of own medications, and ability to handle finances) are summed for a total score ranging from 0 (low function, dependent) to 8 (high function, independent) for women and 0 (low function, dependent) to 5 (high function, independent) for men
Everyday Problem Solving Skills | Day 1
  Everyday Problems Test is a 42 iteme measure of everyday function in several categories (consumerism, meal preparation, medication use, financial management, transportation, phone usage, and housekeeping). Categorical scores are summed to calculate a total score ranging from 0 - 42 with greater scores indicating better everyday problems solving skills.
Depression | Day 1
  Patient Health Questionnaire - 9 is a measure of depressive symptoms, 9-items are summed for a total score ranging from 0-27 with higher scores indicating more severe depressive symptoms
Health Related Quality of Life | Day 1
  Medical Outcomes Study - HIV is a 35-item questionnaire with subscales (health perceptions, pain, physical functioning, role functioning, social functioning, cognitive functioning, mental health, energy, health distress, quality of life, and health transition. Subscales are summed for a total score between 0 and 100 with higher scores indicating better health or well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Shameka L Cody, PhD, Principal Investigator — The University of Alabama
Locations (1):
- University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No